CLINICAL TRIAL: NCT04658940
Title: AcQBlate Force Sensing Ablation System US IDE for Atrial Flutter (AcQForce Flutter)
Acronym: AcQForce AFL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Acutus Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-21; CLP-21-EU (Other: Acutus Medical, Inc.); NCT04657055 (obsolete NCT alias)
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Typical Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Non-randomized (Experimental): All subjects with typical atrial flutter will undergo percutaneous catheter ablation of the cavotricuspid isthmus using the AcQBlate Force Sensing System.
  Interventions: Device: AcQBlate® Force Sensing Ablation System

INTERVENTIONS:
Device: AcQBlate® Force Sensing Ablation System — Percutaneous catheter ablation of the cavotricuspid isthmus
  Other Names: AcQBlate Force Sensing System; AcQBlate Force

SUMMARY:
The Acutus Medical AcQForce Flutter clinical study is a prospective, multi-center, non-randomized global study designed to demonstrate the safety and effectiveness of the AcQBlate Force Sensing Ablation System in the ablation management of symptomatic cavotricuspid isthmus dependent atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are clinically indicated for de novo catheter ablation of typical atrial flutter.
2. At least one (1) documented episode of typical atrial flutter within 180 days (6 months) prior to enrollment, documented by 12-lead ECG.
3. Age 18 years or older at time of consent.
4. Subjects are willing and able to provide written informed consent to participate in the study and agree to comply with all follow-up visits and evaluations.

Exclusion Criteria:

1. In the opinion of the Investigator, any contraindication to the planned atrial ablation, including contraindications to anticoagulation therapy and any other significant uncontrolled or unstable medical condition (e.g. sepsis, acute metabolic illness, chronic kidney disease).
2. Inability to entrain CTI dependent AFL by standard pacing at procedure.
3. Any prior right atrial cavotricuspid isthmus ablation.
4. Any cardiac ablation for non-atrial flutter arrhythmias within 90 days prior to enrollment.
5. Any patient scheduled or anticipating an AF ablation within the follow-up period.
6. Use of amiodarone within 120 days prior to procedure.
7. Cardiac surgery within 60 days prior to enrollment.
8. ST-elevation myocardial infarction (STEMI) within 60 days prior to enrollment
9. Current unstable angina.
10. Documented atrial or ventricular tumors, clots, thrombus, within 30-days prior to enrollment.
11. Any history of a known hematologic disorder (bleeding/clotting).
12. Implantation of permanent leads of an implantable device in or through the right atrium within 90-days prior to enrollment.
13. Subjects with New York Heart Association (NYHA) Class IV heart failure within 6-months prior to enrollment.
14. Subjects with an ejection fraction less than 30% within 90 days of enrollment.
15. Percutaneous Transluminal Coronary Angioplasty (PTCA) within 30-days of enrollment.
16. Clinically significant structural heart disease (including moderate to severe tricuspid valve regurgitation, tricuspid valve stenosis, or tricuspid valve replacement; Ebstein's anomaly, or other congenital heart disease) that would preclude catheter introduction and placement, as determined by the Investigator.
17. Any cerebral ischemic/infarct event (excluding transient ischemic attacks) within 180 days prior to enrollment.
18. Body Mass Index (BMI) >42 kg/m2.
19. International Normalized Ratio (INR) > 3.
20. Severe uncontrolled systemic hypertension (systolic pressure > 240 mm Hg) within the last 30-days.
21. Women who are pregnant or plan to become pregnant within the course of their participation in the investigation.
22. Current enrollment in any other study protocol where testing or results from the study may interfere with the procedure or outcome measurements for this study.
23. Any other condition that, in the judgment of the Investigator, makes the patient a poor candidate for this procedure, the study or compliance with the protocol (includes vulnerable patient population, mental illness, addictive disease, terminal illness with a life expectancy of less than two years, extensive travel away from the research center).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-06-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- United States (20):
  - AZ Cardiovascular Research Center, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - John Muir Health, Concord, California
  - San Diego Cardiac Center Medical Group, Inc., San Diego, California
  - Hartford Hospital, Hartford, Connecticut
  - BayCare Heath, Clearwater, Florida
  - Celebration Hospital, Orlando, Florida
  - Bayfront Health, St. Petersburg, Florida
  - St Alphonsus Health System, Boise, Idaho
  - Kansas City Heart Rhythm Institute, Overland Park, Kansas
  - Baptist Lexington Medical Center, Lexington, Kentucky
  - MedStar Health Research Institute, Hyattsville, Maryland
  - Adventist Healthcare | White Oak Medical Center, Silver Spring, Maryland
  - Adventist Healthcare, Inc, Silver Spring, Maryland
  - Weill Cornell, New York, New York
  - Ohio State Med Ctr, Columbus, Ohio
  - ProMedica Physician Cardiology, Toledo, Ohio
  - Penn State Health, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
- Belgium (2):
  - ZNA Middelheim, Antwerp
  - Jessa Ziekenhuis, Hasselt
- United Kingdom (2):
  - James Cook University Hospital, Middlesbrough
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject classification:
  Screen Failure: exclusion criteria identified. Enrolled: study eligible by meeting all the inclusion and none of the exclusion criteria, up to the point of the procedure (defined as the AcQBlate® FORCE inserted into the body).
  Attempted: the AcQBlate® FORCE was inserted into the body and not used for RF ablation.
  Treated: the AcQBlate® FORCE was inserted into the body and used for RF ablation.
Groups:
- All Study Participants: All subjects with typical atrial flutter will undergo percutaneous catheter ablation of the cavotricuspid isthmus using the AcQBlate Force Sensing System.
  AcQBlate® Force Sensing Ablation System: Percutaneous catheter ablation of the cavotricuspid isthmus
Period: Overall Study
Arm/Group | All Study Participants
Started | 115
Completed | 114
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 43
  >=65 years | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (10.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 90
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 110
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 107
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 14
  United States | 91
  United Kingdom | 10
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.41 (4.59)

OUTCOME MEASURES:

1. Primary Outcome: Subjects Free From Procedure/Device Related Serious Adverse Events (SAEs)
Description: Subjects free from a composite list of pre-specified procedure/device related Serious Adverse Events (SAEs)
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 115
Participants | 115

2. Primary Outcome: Subjects Achieving Acute Procedural Success
Description: Acute procedural success is defined as the demonstration of bidirectional cavotricuspid isthmus block at least 20 minutes following the last radiofrequency application at the cavotricuspid isthmus with the investigational System.
Time Frame: 20 minutes post ablation
Population: Of the 115 subjects enrolled, 5 were attempted and had the venous access portion of the ablation procedure initiated and the AcQBlate® FORCE was inserted into the body and not used for RF ablation. Of the 110 Treated subjects, one subject was unevaluable (categorized as BDB indeterminant) therefore 109 subjects were included in primary effectiveness endpoint calculations.
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 109
Participants | 102

ADVERSE EVENTS:
Time Frame: 30 days post-procedure
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/115
Serious Adverse Events (participants affected / at risk) | 12/115
Other Adverse Events (participants affected / at risk) | 32/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=115)
Atrioventricular block second degree (Cardiac disorders) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 1 (1)
Chronic left ventricular failure (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Infection (Infections and infestations) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Study Participants (N=115)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (4)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Pericarditis (Cardiac disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Groin abscess (Infections and infestations) | 1 (1)
Incision site erythema (Injury, poisoning and procedural complications) | 1 (1)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 4 (4)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1)
Haematoma (Vascular disorders) | 6 (6)
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT04658940/Prot_SAP_000.pdf